CLINICAL TRIAL: NCT05389618
Title: Dietary Challenges in the Population of Nursing Homes' Residents in Slovenia
Brief Title: Dietary Challenges in the Population of Nursing Homes' Residents
Acronym: NUTRICARE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: National Institute of Public Health, Slovenia (Other Government); University Medical Centre Ljubljana (Other); Slovenian Research Agency (Other)
Responsible Party: Sponsor
Other Study IDs: Z3-3213; KME 0120-531/2021/13 (Other: National Medical Ethics Committee (Slovenia))
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Nutritional Status; Nutrient Deficiency; Micronutrient Deficiency; Vitamin D Deficiency; Vitamin B 12 Deficiency; Folic Acid Deficiency; Iron-deficiency; Protein Deficiency; Sarcopenia; Obesity; Diet
Keywords: dietary intake; nutritional status; micronutrients; Slovenia; Europe
MeSH Terms: conditions — Vitamin D Deficiency; Vitamin B 12 Deficiency; Folic Acid Deficiency; Anemia, Iron-Deficiency; Protein Deficiency; Sarcopenia; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood samples will be freezed for possible further analyses on markers related with nutrition & health
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older adults 65-80 years
  Interventions: Other: Diagnostic Tests
- Older adults above 80 years
  Interventions: Other: Diagnostic Tests

INTERVENTIONS:
Other: Diagnostic Tests — Assessment of socio-demographic parameters, anthropometric and body composition parameters, food intake (dietary recalls, food propensity questionnaire) and nutritional status (blood biomarkers)

SUMMARY:
To obtain up-to-date data on nutritional status of older adults, a national dietary survey will be conducted in 2022/2023, providing data on the consumption of foods and enabling the assessment intakes of energy and specific nutrients. Participating subjects will be also screened for micronutrient status using blood biomarkers (focusing into vitamin D, folic acid, vitamin B12, and iron).

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Has been in the elderly care institution (nursing home) for at least 3 months before joining the study
* Care category: I., II., III.A
* The person can feed independently or with minimal help
* Agrees to be included in the study (signed a statement of consent)

Exclusion Criteria:

* The person has an acute illness
* The person is a dialysis patient
* Temporary special diet / fasting / gastrointestinal cleansing (i.e. due to (pre)planned examinations / procedures)
* The person cannot be weighted by the usual weighing scale or chair weighing scale
* Protégé of the day care center
* Located in the red zone of the elderly care institution (nursing home) (COVID-19 measures)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This observational study is conducted on randomly selected residents of 18 different nursing homes, located in all regions in Republic of Slovenia, using described inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of protein intake | 1 year
  epidemiology of protein intake will be investigated from food records [g/day]
Assessment of energy intake | 1 year
  epidemiology of energy intake will be investigated from food records [kJ/day]

SECONDARY OUTCOMES:
Assessment of inadequate vitamin D status | 1 year
  epidemiology of vitamin D status will be investigated using serum 25-OH-vitamin D concentration
Assessment of inadequate folate status | 1 year
  epidemiology of folate status will be investigated using serum folate concentration
Assessment of inadequate vitamin B12 status | 1 year
  epidemiology of vitamin B12 status will be investigated using serum vitamin B12 concentration
Assessment of inadequate iron status | 1 year
  epidemiology of iron status will be investigated using serum ferritin concentration
Assessment of anemia | 1 year
  epidemiology of anemia will be investigated using serum haemoglobin concentration

OTHER OUTCOMES:
Nutritional intakes | 1 year
  epidemiology of dietary intake of nutrients and fibre will be investigated from food records [g/day]
Body mass index | 1 year
  Weight and height will be combined to report BMI in kg/m^2 and providing insights into prevalence of overweight/obesity
Prevalence of sarcopenia | 1 years
  epidemiology of sarcopenia will be investigated using EWGSOP2 (European Working Group on Sarcopenia in Older People 2) criteria and estimated ASM (apendicular skeletal muscle mass)

CONTACTS AND LOCATIONS:
Overall Officials: Živa Lavriša, PhD, Principal Investigator — Nutrition Institute, Ljubljana; Igor Pravst, PhD, Study Director — Nutrition Institute, Ljubljana; Ivan Eržen, PhD, Study Chair — National Institute of Public Health, Slovenia; Nadan Gregorič, Study Chair — University Medical Centre Ljubljana
Locations (1):
- Nutrition Institute, Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided